CLINICAL TRIAL: NCT04970394
Title: Three-year Prospective Cohort Study of the Effectiveness of Physician Reminders on Cervical Screening Uptake Amongst Non Responders in a UK Primary Care Setting
Brief Title: An Observational Study of GP Verbal Reminders Upon Cervical Screening
Acronym: VRCS
Status: Completed | Type: Observational
Sponsor: Dr. Faizan Awan (Other)
Responsible Party: Sponsor-Investigator, Dr. Faizan Awan, General Practitioner, The Gill Medical Centre
Organization: The Gill Medical Centre (Other)
Other Study IDs: 298846
Record Dates: First submitted 2021-07-11; First posted 2021-07-21 (Actual); Last update posted 2021-08-12 (Actual); Status verified 2021-08

CONDITIONS: HPV-Related Cervical Carcinoma; Physician-Patient Relations
Keywords: Cervical Screening; Primary health care; Physician intervention

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Intervention: The principal investigator reviews the medical notes of all individuals they consult over a period of three years to check if they are non responders. If confirmed as non responder, they receive a three-step verbal intervention:
  1. "Your cervical cancer screening is now overdue."
  2. "The test is easy to perform and saves thousands of lives from cervical cancer every year."
  3. "Should we book an appointment for cervical screening now so that you make sure you have it done?"
     Those who are seen face-to-face receive a fourth intervention:
  4. An appointment slip is given to the patient to hand to the receptionist. This includes the patient's name and the comment, "book an appointment with practice nurse for cervical screening".
  Interventions: Behavioral: Cervical Screening Reminder
- Control: The control group receives standard unstructured reminders regarding their overdue status from any of the 6 other clinicians during appointments and / or reminder letters from the administration team.

INTERVENTIONS:
Behavioral: Cervical Screening Reminder — Verbal reminder and if seen face-to-face, a written appointment booking slip.
  Groups: Intervention

SUMMARY:
Cervical cancer screening is offered to all women in the United Kingdom (UK) between the ages of 24.5 and 64 years of age. The majority of screening is performed in primary care and the rate remains stubbornly below 80%, despite an automated national invitation system. This study is designed to assess the effectiveness of a physician invitation during a telephone or face-to-face primary care appointment upon non responders of automated invitations, to increase the uptake of cervical screening.

DETAILED DESCRIPTION:
It is estimated that between 800 and 2,000 deaths a year are now prevented due to the effectiveness of the UK's national cervical screening programme and mortality rates have dropped by over 75% since the 1970s. These statistics corroborate the importance of the screening programme in reducing mortality from cervical cancer. Cervical screening rates in the UK remains stubbornly below 80% and interventions are needed to attract the 20% who are missing out on screening. This prospective observational study is designed to measure the impact of a physician intervention in a usual healthcare environment, amongst a heterogeneous patient population to yield replicable real-world results. The intervention arm will receive a physician intervention to inform them of their overdue screening status, remind them of the importance of cervical screening and guide them to book a screening appointment. The screening rate in the intervention arm will be compared to a control made up of patients seen by other clinicians and receiving unstructured reminders. The results will assist physicians in deciding whether a structured intervention is anymore effective than the unstructured advice currently given at improving screening rates in the non responder population.

ELIGIBILITY:
Inclusion Criteria:

* Registered patient with a cervix
* Non responder to cervical screening invitation

Exclusion Criteria:

* Incorrectly reminded i. Coding errors ii. Human error
* Temporary patients i. Did not remain registered for minimum of 6 months following intervention
* Screening refusal
* Inappropriate to include i. Terminal illness ii. Prolonged hospitalisation iii. Death due to non-cervical cancer attributable cause

Ages: 25 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Any individual with a cervix
Study Population: Patients registered at the Gill Medical Centre, who have a cervix, are eligible for cervical screening and have been non responders to the automated national invitation. These patients are opportunistically recruited when they are consulted by the principal investigator.
Sampling Method: Probability Sample
Enrollment: 724 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2020-02-29 (Actual); Study Completion 2021-03-03 (Actual)

PRIMARY OUTCOMES:
Uptake of Cervical Screening | Up to 1 year post intervention
  The number of patients who undergo cervical screening

SECONDARY OUTCOMES:
Time to book screening | Up to 1 year post intervention
  Length of time taken to undergo screening following intervention

CONTACTS AND LOCATIONS:
Overall Officials: Faizan A Awan, MBChB MRCGP, Principal Investigator — The Gill Medical Centre
Locations (1):
- The Gill Medical Centre, Salford, Greater Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
The IPD will be shared with researchers who confirm the purpose of their request and are affiliated with a research organisation.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Immediately available for up to 10 years post-publication.
Access Criteria: Contact principal investigator via e-mail.

REFERENCES:
- [Background] Everett T, Bryant A, Griffin MF, Martin-Hirsch PP, Forbes CA, Jepson RG. Interventions targeted at women to encourage the uptake of cervical screening. Cochrane Database Syst Rev. 2011 May 11;2011(5):CD002834. doi: 10.1002/14651858.CD002834.pub2. PMID 21563135